CLINICAL TRIAL: NCT05009732
Title: A Randomized, Double-blind, Placebo-Controlled, Phase III Study to Evaluate the Efficacy and Safety of Proxalutamide (GT0918) in Hospitalized COVID-19 Subjects
Brief Title: A Study to Evaluate the Efficacy and Safety of Proxalutamide (GT0918) in Hospitalized COVID-19 Subjects
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Suzhou Kintor Pharmaceutical Inc, (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GT0918-US-3002
Record Dates: First submitted 2021-08-16; First posted 2021-08-17 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Covid19
Keywords: SARS-CoV-2; Covid
MeSH Terms: conditions — COVID-19 | interventions — proxalutamide; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Proxalutamide (GT0918) plus standard of care (Experimental): Participants receive 300mg once daily orally plus standard of care for 7 days and can be extended up to 14 days per investigator discretion
  Interventions: Drug: GT0918; Drug: Standard of care
- Placebo plus standard of care (Placebo Comparator): Participants will receive placebo tablets matching Proxalutamide (GT0918) orally plus standard of care for 7 days and can be extended up to 14 days per investigator discretion
  Interventions: Drug: Standard of care; Drug: Matching placebo

INTERVENTIONS:
Drug: GT0918 — 300mg once daily orally
  Other Names: Proxalutamide
  Arms: Proxalutamide (GT0918) plus standard of care
Drug: Standard of care — Local standard of care per written policies or guidelines
  Other Names: SoC
Drug: Matching placebo — Matching placebo
  Other Names: Placebo
  Arms: Placebo plus standard of care

SUMMARY:
This study is an adaptive Phase III randomized double-blind placebo-controlled trial to evaluate the efficacy and safety of Proxalutamide (GT0918) in hospitalized adults diagnosed with COVID-19. The study is a multicenter trial that will be conducted globally. The study will compare GT0918 plus standard of care (SOC) with the placebo plus SOC. Approximately 762 subjects will be randomized in a 1:1 ratio to either GT0918 plus SOC or placebo plus SOC group.

DETAILED DESCRIPTION:
Coronavirus disease 2019 (COVID-19) emerged in late 2019 and spread rapidly, resulting in a global pandemic.SARS-CoV-2 encodes nonstructural and structural proteins required for its viral life cycle. Among them, the spike glycoprotein plays a pivotal role in SARS-CoV-2 infection by recognizing and attaching to ACE2 transmembrane protein on host cells. Kintor protocol has been designed to evaluate efficacy and safety of GT0918 in hospitalized subjects with COVID-19 illness. The target population of this study are hospitalized subjects with COVID-19 illness with positive SARS-CoV-2 virus test within 72 hours of randomization. The study will evaluate anti-androgen therapy may effectively prevent progression to the more severe form of COVID-19 illness and death, shorten the time to sustained recovery and decrease the mortality rate. Subject will receive either GT0918 plus standard of care or matched placebo plus standard of care. GT0918/placebo will be given 300mg orally once a day around 30 minutes after meal for 7 days and can be extended up to 14 days per investigator discretion

ELIGIBILITY:
Inclusion Criteria:

1. Subject (or legally authorized representative) provides informed consent prior to initiation of any study procedures.
2. Subject (or legally authorized representative) understands and agrees to comply with planned study procedures.
3. Male and non-pregnant female subjects with age ≥18 years of age at the time of randomization.
4. Admitted to a hospital with symptoms suggestive of severe COVID-19.
5. Has laboratory-confirmed SARS-CoV-2 infection as determined by PCR or other commercial or public health assay (including rapid antigen test) in any specimen, as documented by either of the following:

   * PCR positive in sample collected < 72 hours prior to randomization; OR
   * PCR positive in sample collected ≥ 72 hours prior to randomization, documented inability to obtain a repeat sample (e.g. due to lack of testing supplies, limited testing capacity, results taking > 24 hours, etc) AND progressive disease suggestive of ongoing SARS-CoV-2 infection.
6. Illness of any duration, and at least one of the following:

   * Shortness of breath, RR≥30 /minute
   * Clinical signs indicative of progressive aggravation, lung radiographic infiltrates by imaging (chest x-ray, CT scan, etc.) showing >50% progression within 24-48 hours
   * PaO2/FiO≤300mmHg 1mmHg=0.133kPa
   * Resting state SpO2 ≤ 93% on room air
7. All women of childbearing potential defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) and is not postmenopausal. Highly effective contraception methods include:

   * Total Abstinence (when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception, or
   * Use of one of the following combinations (a+b or a+c or b+c):

     1. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception.
     2. Placement of an intrauterine device (IUD) or intrauterine system (IUS);
     3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository;
   * Female sterilization (have had prior surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment;
   * Male sterilization (at least 6 months prior to screening). For female subjects on the study, the vasectomized male partner should be the sole partner for that subject;
   * In case of use of oral contraception women should have been stable for a minimum of 3 months before taking study treatment. Women are considered post-menopausal and not of childbearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment, is she considered not of childbearing potential;
8. Regardless of their fertility status, male subjects must agree to either remain abstinent (if this is their preferred and usual lifestyle) or use condoms as well as one additional highly effective method of contraception (less than 1% failure rate) or effective method of contraception with nonpregnant women of childbearing potential partners for the duration of the study and until 90 days after the last dose. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.
9. Agree not to participate in another clinical trial for the treatment of COVID-19 through Day 60 after first dose.

Exclusion Criteria:

Subjects are excluded from the study if any of the following criteria apply:

1. ALT/AST > 3 times the upper limit of normal.
2. Serum total bilirubin > 1.5 x ULN (upper limit of normal)
3. Estimated glomerular filtration rate (eGFR) < 30 ml/min (including patients receiving hemodialysis or hemofiltration).
4. Subjects with significant cardiovascular disease as following:

   i. heart failure NYHA class ≥3 ii. left ventricular ejection fraction <50% iii. those with a history of cardiac arrhythmias, including long QT syndrome.
5. Neutropenia (absolute neutrophil count <1000 cells/μL) (<1.0 x 10^3/μL).
6. Lymphopenia (absolute lymphocyte count <200 cells/μL) (<0.20 x 10^3/μL)
7. Pregnancy or breast feeding
8. Anticipated discharge from the hospital or transfer to another hospital which is not a study site within 72 hours.
9. Allergy to any study medication.
10. Received monoclonal antibody, convalescent plasma, or intravenous immunoglobulin [IVIg]) for COVID-19 withing 14 days of screening.
11. Suspected serious, active bacterial, fungal, viral, or other infection (besides COVID-19) that in the opinion of the investigator could constitute a risk when taking investigational product.
12. Have a history of VTE (deep vein thrombosis [DVT] or pulmonary embolism [PE]) within 12 weeks prior to screening or have a history of recurrent (>1) VTE (DVT/PE).
13. Subject taking or had taken an anti-androgen of any type including androgen depravation therapy, 5-alpha reductase inhibitors, etc. within 3 months before dosing.
14. Have participated, within the last 30 days before dosing, in a clinical study involving an investigational intervention. If the previous investigational intervention has a long half-life, 5 half-lives or 30 days, whichever is longer, should have passed.
15. Subjects with active myopathy
16. Is admitted to Intensive Care Units at randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-07-14 (Actual)

PRIMARY OUTCOMES:
The time to Clinical deterioration is evaluated by Day 30. | 30 days from enrollment
  Clinical deterioration is defined as the need for intensive care unit level care (ICU) or invasive mechanical ventilation/ECMO or all-cause mortality by Day 30.

SECONDARY OUTCOMES:
60-day mortality | 60 days from enrollment
  All cause mortality at 60 days after enrollment

CONTACTS AND LOCATIONS:
Locations (30):
- United States (8):
  - Alternative Research Associates LLC., Hialeah, Florida
  - Sparrow Hospital, Lansing, Michigan
  - Hannibal Clinic (HC), Hannibal, Missouri
  - Raymond G. Murphy VA Medical Center, Albuquerque, New Mexico
  - Saint Lawrence Health System, New York, New York
  - Ascension St. John Medical Center, Tulsa, Oklahoma
  - Medical City Fort Worth, Fort Worth, Texas
  - PRX Research, Mesquite, Texas
- China (3):
  - Shanghai Public Health Clinical Center, Zhujing, Shanghai Municipality
  - The Third People's Hospital of Shenzhen, Longgang District, Shenzhen
  - Beijing Ditan Hospital Capital Medical University, Beijing
- Philippines (6):
  - Davao Doctors Hospital, Davao City, Davao Region
  - St. Paul's Hospital, Iloilo City, Iloilo
  - Philippine General Hospital, Malina, Metro Malina
  - Mary Johnston Hospital (MJH), Manila, National Capital Region
  - Quirino Memorial Medical Center, Quezon City, National Capital Region
  - Lung Center of the Philippines, Quezon City
- South Africa (6):
  - Johese Clinical Research: Unitas, Centurion
  - Drs Sarvan and Moodley, Durban
  - TASK Eden, George
  - Johese Clinical Research ZAH, Pretoria
  - Dr JM Engelbrecht Practice, Vergelegen Mediclinic, Somerset
  - Clinical Projects Research, Worcester
- Ukraine (7):
  - Communal Noncommercial Profit, Dnipro, Dnipro Oblast
  - Ivano-Frankivsk Clinical Regional Infectious Diseases Hospital, Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Kharkiv city clinical hospital #13, Kharkiv, Kharkivs’ka Oblast’
  - CNE of Kharkov RC Reg Cl Infectious Hospital, Kharkiv, Kharkivs’ka Oblast’
  - City Clinical infectious Hospital, Odesa, Odesa Oblast
  - Poltava Regional Clinical, Poltava, Poltava Oblast
  - CCH #1 Vinnytsia M.I.Pyrogov NMU Ch of Infectious Diseases, Vinnytsia, Vinnytsia Oblast

IPD SHARING:
Plan to Share IPD: No